## Effects of Simethicone and Multilac Baby in Infantile Colic

| <b>24-hours Parents Da</b><br>Name:<br>Date: | ay Repo | | Date | of bir | rth: | | <br> | | | Page-No.: | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Night | 2 | 3 | 4 | Morning<br>4 5 6 7 | 8 | 9 | 10 | 11 | Afternoon<br>12 13 14 | 16 | 17 | Evenr<br>17 18 19 | 21 | 22 23 24 |
| Sleeping | | | | | | | | 10 | | 12 | | 17 | | | |
| Restlessness /<br>whining | | | | | | | | | | | | | | | |
| - Duration (min) | | | | | | | | | | | | | | | |
| Crying | | | | | | | | | | | | | | | |
| - Duration (min) | | | | | | | | | | | | | | | |
| Breastfeeding | | | | | | | | | | | | | | | |
| Formula feeding | | | | | | | | | | | | | | | |
| Administration of treatment | | | | | | | | | | | | | | | |
| Comments | | | | | | | | | | | | | | | |